CLINICAL TRIAL: NCT00967733
Title: Effect of Alpha-Linolenic Acid on Blood Markers of Inflammation
Brief Title: Alpha-Linolenic Acid and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: P-16261-101
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- High ALA-Low Linoleic (Active Comparator)
  Interventions: Dietary Supplement: Flaxseed oil-Olive oil
- Low ALA-Low Linoleic (Placebo Comparator)
  Interventions: Dietary Supplement: Olive oil-olive oil
- High ALA-High Linoleic (Active Comparator)
  Interventions: Dietary Supplement: Flaxseed oil-sunflower oil
- Low ALA-High Linoleic (Placebo Comparator)
  Interventions: Dietary Supplement: Olive oil-sunflower oil

INTERVENTIONS:
Dietary Supplement: Flaxseed oil-Olive oil — 2 or 4 gr per day alpha-linolenic acid pill and olive oil used for cooking
  Arms: High ALA-Low Linoleic
Dietary Supplement: Olive oil-olive oil — 1 gr olive oil pill and olive oil used for cooking
  Arms: Low ALA-Low Linoleic
Dietary Supplement: Flaxseed oil-sunflower oil — 2 or 4 gr per day alpha linolenic acid pill and sunflower oil used for cooking
  Arms: High ALA-High Linoleic
Dietary Supplement: Olive oil-sunflower oil — 1 gr olive oil pill and sunflower oil used for cooking
  Arms: Low ALA-High Linoleic

SUMMARY:
The optimal type of oil to prevent cardiovascular disease (CVD) is uncertain. In general, unsaturated oils with higher content of cis-monounsaturated fatty acids (MONO) or cis-polyunsaturated fatty acids (PUFA) are preferable over those rich in saturated fatty acids. However, unsaturated oils can vary in their relative contents of n-6 and n-3 fatty acids (specifically alpha-linolenic acid (ALA)). Some investigators advocate that oils rich in ALA are cardioprotective, while others suggest that optimal cardioprotective effects can only be obtained when oils are lower in n-6 fatty acids (mainly linoleic acid) in addition to being higher in ALA. It is hypothesized that increased ALA would result in beneficial effects on inflammatory markers. The objective of this trial is to establish definitively the biological effects of ALA with and without reductions in linoleic acid on inflammatory markers linked to CVD.

DETAILED DESCRIPTION:
This study is a dietary trial that examines the effects of increasing ALA by 2 gr or 4 gr per day, with and without decreasing linoleic acid, on inflammatory markers linked to CVD. Trial participants (n=136), approximately 50% women, 50% men) are age 50 and older and living in the town of Montana, Bulgaria during the study. The study uses a double-blinded placebo-controlled, randomized cross-over design. Combinations of two oils that are considered healthy (sunflower and olive) and an ALA supplement containing either 2 or 4 gr of ALA (supplied as flaxseed oil) or placebo are consumed for 6 weeks each: sunflower-ALA (high linoleic-low ALA), sunflower-placebo (high linoleic-low ALA), olive-ALA (low-linoleic-high ALA) and olive-placebo (low linoleic-low ALA). The participants are indicated to keep their usual diet and physical activity through-out the study. The primary endpoints are plasma levels of inflammatory markers. Secondary endpoints include systolic and diastolic blood pressure, and plasma levels of LDL cholesterol, HDL cholesterol and triglycerides.

SPECIFIC AIMS

To determine the effect of increasing ALA by 2 or 4 gr per day in the context of a diet that that is high in linoleic acid (~13% energy) on inflammatory markers. The ALA effect will be tested by comparing ALA supplement vs. placebo while using sunflower oil for cooking at home. We hypothesize that ALA has favorable effects on inflammatory markers in the context of a diet that is high in linoleic acid.

To determine the effect of increasing ALA by 2 or 4 gr per day in the context of a diet that that is low in linoleic acid (~6% energy) on inflammatory markers. The ALA effect will be tested by comparing ALA supplement vs. placebo while using olive oil for cooking at home. We hypothesize that ALA has favorable effects on inflammatory markers in the context of a diet that is low in linoleic acid.

SECONDARY AIMS

To determine the effect of reducing linoleic acid from a high level (~13% energy) to a low level (~6% energy) while keeping ALA at a high level (2 or 4 gr per day) on plasma levels of inflammatory markers. The reduction in linoleic acid will be tested by comparing sunflower to olive oil while taking the ALA supplement. We hypothesize that reducing linoleic acid does not affect inflammatory markers when ALA intake is high.

To determine the effect of reducing linoleic acid from a high level (~13% energy) to a low level (~6% energy) while keeping ALA at a low level (placebo) on plasma levels of inflammatory markers. The reduction in linoleic acid will be tested by comparing sunflower to olive oil while taking the placebo. We hypothesize that reducing linoleic acid does not affect inflammatory markers when ALA intake is low.

To determine whether the intervention contrasts specified in the specific aims and secondary aims 1 & 2 affect plasma levels of LDL cholesterol, HDL cholesterol and triglycerides and blood pressure.

We hypothesize that ALA has favorable effects on plasma triglycerides and blood pressure compared to placebo regardless of whether linoleic acid is high or low.

We hypothesize that lowering linoleic acid has favorable effects on plasma HDL cholesterol but unfavorable effects on LDL cholesterol,regardless of whether ALA is high or low.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older at time of enrollment
* Willing to cook and eat foods prepared exclusively with the study oils and nothing else every day of the week at least 2 meals per day for 24 weeks
* Willing to eat no more than one meal per week prepared out of the home
* Willingness to take 4 or 8 capsules with ALA or placebo every day for 24 weeks
* Willingness to provide personal and next of kin address and phone number for follow-up visits to the home.
* Willingness to complete measurement procedures and blood draws.
* Ability and willingness to provide informed consent to be screened and to take part of the study.

Exclusion Criteria:

Medication Exclusions

• Unstable dose of medications during the past 2 months that raise or lower blood pressure, lipids or glucose. Unstable dose is a dose change in the past 6 months or less than 6 months of treatment.

Medical History Exclusions

* Active or prior CVD (stroke, MI, PTCA, CABG, congestive heart failure, symptomatic ischemic heart disease (angina), or CVD-related therapeutic procedure).
* Cancer diagnosis or treatment in past two years (however, persons with non-melanoma skin cancer, localized breast cancer, or localized prostate cancer can enroll if they did not require systemic chemotherapy)
* Active inflammatory bowel disease, malabsorption, or major GI resection
* Chronic renal disease
* Any serious illness not otherwise specified that would interfere with participation
* Stage 2 hypertension (SBP > 160 or DBP > 100 mmHg) based on the mean of 3 measurements on the screening visit, as well as a systolic BP > 170 or diastolic BP > 105 at any of the measurements

Other Exclusions

* Eat fish more than once per week including canned fish
* Significant oil preferences, intolerances, dietary habits, or dietary requirements that would interfere with adherence
* Planning to leave the area for more than two weeks prior to the anticipated end of participation
* Current participation in another study that manipulates diet or that will affect the outcome of this study
* Taking vitamin, vegetable oil, fish-oil, weight-loss, soy, mineral, or herbal supplements that cannot be stopped
* Unable to measure blood pressure (due to arm circumference > 50 cm)
* Investigator judgment (e.g. for concerns over adherence, or follow-up or for inappropriate behavior)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Markers of inflammation | 6 weeks

SECONDARY OUTCOMES:
Plasma lipids and blood pressure | 6 weeks